CLINICAL TRIAL: NCT01219231
Title: Exercise in Elderly Individuals With Impaired Glucose Tolerance: Beneficial for Vasculature and Neurons?
Brief Title: Effects of Physical Activity on the Brain in Impaired Glucose Tolerance (IGT)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Principal Investigator, Agnes Flöel, Prof, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: exercise_neuromod
Record Dates: First submitted 2010-10-12; First posted 2010-10-13 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Impaired Glucose Tolerance
Keywords: Exercise; elderly; cognition; prevention; cognitive decline; Lifestyle
MeSH Terms: conditions — Glucose Intolerance; Motor Activity; Cognitive Dysfunction | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise (Experimental)
  Interventions: Behavioral: Exercise
- Placebo (Placebo Comparator)
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — 6 months of aerobic exercise

SUMMARY:
The researchers will investigate whether exercise could provide positive effects on general brain functions in elderly people with impaired glucose tolerance.

DETAILED DESCRIPTION:
The age-related degradation of cognitive functions even to the point of neurodegenerative disorders such as Alzheimer's disease are a growing public-health concern with devastating effects.

Referring to animal data, empirical studies, and pilot human trials, exercise should improve cognitive functions such as learning and memory. To test this hypothesis, the researchers study general brain functions in elderly subjects (50-80 years old) with impaired glucose tolerance during a short term exercise program.

ELIGIBILITY:
Inclusion Criteria:

* subjects with impaired glucose tolerance
* 50-65 years old
* moderate to heavy weight (BMI 25-35)
* must be able to do exercise intervention

Exclusion Criteria:

* diabetes
* younger than 50 years
* BMI < 25
* psychiatric medication
* severe disease
* MMSE < 26
* severe cardiovascular disorders

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2010-08; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Auditory Verbal Learning Task | Prior to intervention and after 6 months of intervention

SECONDARY OUTCOMES:
Functional/Structural brain changes | Prior to intervention and after 6 months of intervention
Plasma biomarkers | Prior to intervention and after 6 months of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Flöel, MD, Prof., Principal Investigator — Charité University Berlin
Locations (1):
- Department of Neurology, Charité Universitätsmedizin, Berlin, State of Berlin, Germany